CLINICAL TRIAL: NCT05337358
Title: Clinical Performance of Fiber Reinforced FRC Base and Bonded CAD/CAM Resin Composite Endocrowns Versus Conventional Lithium Disilicate Endocrowns in Posterior Teeth (1y Randomized Clinical Trial).
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sameh Abou-steit, Lecturer of fixed prosthodontics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-2021-3-040
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Clinical Performance
Keywords: Lithium dislocate; fiber reinforced composite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lithium disilicate (Active Comparator): The intervention will be: Prosthetic endocrown
  Interventions: Procedure: endocrown
- Fiber reinforced composite (Active Comparator): The intervention will be: Prosthetic endocrown
  Interventions: Procedure: endocrown

INTERVENTIONS:
Procedure: endocrown — endocrown

SUMMARY:
In patients with endodontically treated molar teeth indicated for endocrown, will the fiber reinforced FRC base and bonded CAD/CAM resin composite endocrowns restorations have a similar clinical performance to the conventional lithium disilicate endocrown over one year?

ELIGIBILITY:
Inclusion Criteria:

* Patients with good oral hygiene
* Patients having one or more endodontically treated molars that need prosthetic restoration.
* Molars should have enough tooth structure for endocrown restoration with minimum 3 walls with thickness not less than 1.5 mm and gingival step placed supragingival
* Fully erupted molars
* Molars free of developmental defect
* Healthy periodontium
* Absence of periapical pathosis
* Acceptable endodontic treatment and proper bone support

Exclusion Criteria:

* Patients with bad oral hygiene
* Patients with active periodontal disease
* Patients with missing teeth opposing to the area intended for restoration
* Patients with parafunctional habits or psychiatric problems or unrealistic expectation.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-04-11 (Estimated); Study Completion 2023-04-11 (Estimated)

PRIMARY OUTCOMES:
clinical performance | 2 years
  Using the modified United States Public Health Service criteria (Modified USPHS)- categorical

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Sh Abou-steit, PhD, Principal Investigator — Lecturer of Fixed Prosthodontics
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided